CLINICAL TRIAL: NCT04902040
Title: An Open-label, Single-Center, Phase 1b/2 Study to Evaluate the Safety of Plinabulin in Combination With Radiation/Immunotherapy in Patients With Select Advanced Malignancies After Progression on PD-1 or PD-L1 Targeted Antibodies
Brief Title: Plinabulin in Combination With Radiation/Immunotherapy in Patients With Select Advanced Cancers After Progression on PD-1 or PD-L1 Targeted Antibodies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI requested.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0296; NCI-2021-03489 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0296 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-05; First posted 2021-05-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: Advanced Bladder Carcinoma; Advanced Lung Non-Small Cell Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Melanoma; Advanced Merkel Cell Carcinoma; Advanced Renal Cell Carcinoma; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage III Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Clinical Stage IV Merkel Cell Carcinoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage III Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Pathologic Stage IV Merkel Cell Carcinoma AJCC v8; Stage III Bladder Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Bladder Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IVA Bladder Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Bladder Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms; Lung Neoplasms; Carcinoma, Renal Cell | interventions — atezolizumab; avelumab; durvalumab; Immunoglobulin G; Disulfides; Nivolumab; pembrolizumab; NPI 2358; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (radiation therapy, plinabulin, immunotherapy) (Experimental): Patients undergo radiation therapy on days 1-3, 1-4, or 1-5 of cycle 1. Patients may undergo additional radiation in cycle 2 at the discretion of treating physician. Patients receive plinabulin IV over 30-60 minutes on days 1 and 4 of cycle 1, days 1 and 4 of cycle 2 (if receiving radiation therapy in cycle 2), and day 1 and or 15 (any day receiving immunotherapy) of subsequent cycles. Patients also receive immunotherapy consisting of either: avelumab IV over 1 hour on days 1 and 15; atezolizumab over 30-60 minutes on day 1; durvalumab IV over 1 hour on days 1 and 15; nivolumab IV over 30-60 min on days 1 and 15; or pembrolizumab IV over 30 min on day 1. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Avelumab; Biological: Durvalumab; Biological: Nivolumab; Biological: Pembrolizumab; Drug: Plinabulin; Radiation: Radiation Therapy
- Arm B (radiation therapy, immunotherapy) (Active Comparator): Patients undergo radiation therapy on days 1-3, 1-4, or 1-5 of cycle 1. Patients may undergo additional radiation in cycle 2 at the discretion of treating physician. Patients also receive immunotherapy consisting of either: avelumab IV over 1 hour on days 1 and 15; atezolizumab over 30-60 minutes on day 1; durvalumab IV over 1 hour on days 1 and 15; nivolumab IV over 30-60 min on days 1 and 15; or pembrolizumab IV over 30 min on day 1. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Avelumab; Biological: Durvalumab; Biological: Nivolumab; Biological: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Plinabulin — Given IV
  Other Names: NPI-2358
  Arms: Arm A (radiation therapy, plinabulin, immunotherapy)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of plinabulin in combination with radiation therapy and immunotherapy in patients with select cancers that have spread to other places in the body (advanced) after progression on PD-1 or PD-L1 targeted antibodies. Plinabulin blocks tumor growth by targeting both new and existing blood vessels going to the tumor as well as killing tumor cells. Immunotherapy may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving plinabulin in combination with radiation therapy and immunotherapy may work better in treating advanced cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of plinabulin when administered in combination with radiation/immunotherapy regimen in subjects with select advanced solid malignancies after progression on anti-PD-1/PD-L1 monoclonal antibody (mAb).

II. To assess the objective tumor response rate (complete response + partial response).

SECONDARY OBJECTIVES:

I. To assess disease control rate (complete response, partial response + stable disease).

II. To determine progression-free survival (PFS). III. To assess overall survival.

EXPLORATORY OBJECTIVES:

I. To analyze the gene mutation density within each sample. II. To assess T-cell receptor (TCR) sequencing in tumor tissue and peripheral blood, pre- and post- treatment.

III. To perform imaging mass flow cytometry (CyTOF) and/or single cell ribonucleic acid sequencing (RNAseq) analysis on tumor tissue: Immune phenotyping, including dendritic cell (DC), T cells, tumor-associated macrophage (TAM)s, pre and post treatment.

IV. To conduct phenotyping analysis of immune cells from peripheral blood using multicolor flow cytometry.

V. To evaluate dendritic cell activation from whole blood upon the treatment. VI. To explore general predictive and response biomarker measurements from the collected biomarkers.

OUTLINE: This is a phase Ib, dose-escalation study of plinabulin followed by a phase II study. Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo radiation therapy on days 1-3, 1-4, or 1-5 of cycle 1. Patients may undergo additional radiation in cycle 2 at the discretion of treating physician. Patients receive plinabulin intravenously (IV) over 30-60 minutes on days 1 and 4 of cycle 1, days 1 and 4 of cycle 2 (if receiving radiation therapy in cycle 2), and day 1 and or 15 (any day receiving immunotherapy) of subsequent cycles. Patients also receive immunotherapy consisting of either: avelumab IV over 1 hour on days 1 and 15; atezolizumab over 30-60 minutes on day 1; durvalumab IV over 1 hour on days 1 and 15; nivolumab IV over 30-60 min on days 1 and 15; or pembrolizumab IV over 30 min on day 1. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo radiation therapy on days 1-3, 1-4, or 1-5 of cycle 1. Patients may undergo additional radiation in cycle 2 at the discretion of treating physician. Patients also receive immunotherapy consisting of either: avelumab IV over 1 hour on days 1 and 15; atezolizumab over 30-60 minutes on day 1; durvalumab IV over 1 hour on days 1 and 15; nivolumab IV over 30-60 min on days 1 and 15; or pembrolizumab IV over 30 min on day 1. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have one of seven histologically or cytologically confirmed malignant neoplasms (non-small cell lung cancer, small cell lung cancer, renal cell cancer, bladder cancer, Merkle cell cancer, microsatellite instability high (MSI-H) cancer (any histology), and melanoma) progressed on previous anti-PD-1/PD-L1 mAb treatment +/- chemotherapy or anti-CTLA4 requiring further treatment
* At least one lesion is amenable to radiation
* At least one additional non-contiguous lesion that has not been irradiated amenable to radiographic evaluation
* Have measurable disease based on immune-related response criteria (immune-related Response Evaluation Criteria In Solid Tumors [RECIST])
* Tissue must be newly obtained as a core needle biopsy (not fine-needle aspiration [FNA]) of the lesion being evaluated
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subjects must be recovered from any prior major surgery. The major surgery must be performed at least 4 weeks prior to consent date
* Platelets >= 100 x 10^9/L

  * Transfusions and growth factors are allowed
* Hemoglobin >= 9 g/dL

  * Transfusions and growth factors are allowed
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L

  * Transfusions and growth factors are allowed
* White blood cell (WBC) >= 3 x 10^9/L

  * Transfusions and growth factors are allowed
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) (=< 1.5 x ULN if alkaline phosphatase is > 2.5 x ULN) (In the expansion cohort, subjects with known liver involvement may have ALT =< 5 x ULN)
* Alkaline phosphatase < 4 x ULN
* Total bilirubin =< 1 x ULN (In the expansion cohort, subjects with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of =< 3 x ULN)
* Albumin >= 3 g/dL
* Renal function defined as a calculated or measured glomerular filtration rate (GFR) >= 30 mL/min and Cockcroft-Gault equation
* The patient has recovered to grade =< 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies, with the exception of alopecia. The exceptions for such effects are allowed lab values of =< grade 2 specified elsewhere in these inclusion criteria
* Subjects must give informed consent according to the rules and regulations of the individual participating sites
* Negative urine pregnancy test in women of child bearing potential within 7 days of first dose of treatment and subjects of child-bearing potential must agree to use effective contraception during and for 5 months following the last dose of atezolizumab or nivolumab, and for 4 months after the last dose of pembrolizumab, and for 3 months after last dose of durvalumab and avelumab, and for 3 months after your last dose of plinabulin. A woman of childbearing potential is defined as a premenopausal female capable of becoming pregnant. This includes women on oral, injectable or mechanical contraception; women who are single and women whose male sexual partners have been vasectomized or whose male sexual partners have received or are utilizing mechanical contraceptive devices

Exclusion Criteria:

* Evidence of complete or partial bowel obstruction
* Subjects with primary central nervous system (CNS) tumor or CNS tumor involvement. However, subjects with metastatic CNS tumors may participate in this study if the patient is:

  * > 4 weeks from prior therapy completion
  * Clinically stable with respect to the CNS tumor at the time of study entry
  * Not receiving steroid therapy in treating CNS tumor or CNS tumor involvement
  * Not receiving anti-convulsive medications (that were started for brain metastases)
* Need of total parenteral nutrition
* Allergic to any of anti-PD-1/PD-L1 monoclonal antibody (mAb) intended to receive
* Prior exposure to plinabulin
* Pregnancy or lactation
* Radiation (except planned or ongoing palliative radiation to bone outside of the region of measurable disease) =< 3 weeks prior to study drug administration date
* Chemotherapy, or immunotherapy or any other systemic anticancer therapy =< 3 weeks prior to study drug administration date except anti-PD-1/PD-L1 mAb mono or combination therapy
* Diagnosis or recurrence of invasive cancer other than the present cancer within 3 years (except basal or squamous cell carcinoma of the skin that has been definitively treated)
* Major surgery within four weeks before consent date
* Unstable cardiovascular function or active cardiac disease:

  * Symptomatic ischemia (chest pain of cardiac origin),or
  * Uncontrolled clinically significant conduction abnormalities (e.g. ventricular tachycardia on antiarrhythmics are excluded; 1st degree AV block or asymptomatic Left anterior fascicular block (LAFB)/ right bundle branch block (RBBB) will not be excluded),or
  * Congestive heart failure (CHF) of New York Heart Association (NYHA) class >= 3, or
  * Myocardial infarction (MI) within 3 months of consent date
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to the first dose. Active infection with concurrent treatment is acceptable only if the patient is clinically stable
* Subject is known to be positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Significantly diseased (as determined by the PI or treating physician) or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea. Presence of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility
* Treatment with an investigational anti-cancer study drug within 3 weeks prior to study drug administration date
* Concurrent therapy with approved or investigational anticancer therapeutics
* Medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Men whose partner is a woman of child-bearing potential, (i.e. biologically able to conceive), and who is not employing two forms of highly effective contraception. Highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 5 months following the last dose of atezolizumab or nivolumab, for 4 months after the last dose of pembrolizumab, and for 3 months after last dose of durvalumab and avelumab, and for 3 months after your last dose of plinabulin. Women of child-bearing potential is defined as sexually mature women who are not surgically sterile or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of plinabulin
  AEs will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Objective tumor response rate (ORR) (complete response + partial response) | Up to 4 years
  Radiologic evaluations will be performed at screening and every 9 weeks (± 1 week) for 27 weeks (during Q3W dosing) or every 8 weeks (± 1 week) for 24 weeks (during Q4W dosing), then every 12 weeks during treatment cycles in the Treatment Phase regardless of treatment cycles and follow up period. Categorization of response will be based on both immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) and modified Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Disease control rate (complete response, partial response + stable disease) | Up to 4 years
  Assessed according to irRECIST criteria.
Progression-free survival | From the first study dose date to the date of first documentation of confirmed disease progression or death (whichever occurs first), assessed up to 4 years
  Will be analyzed using Kaplan-Meier method or Cox regression.
Overall survival | From the start date of the treatment period until date of death from any cause, assessed up to 4 years
  Will be analyzed using Kaplan-Meier method or Cox regression.

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04902040/ICF_000.pdf